CLINICAL TRIAL: NCT03230045
Title: Effect of Dual Acupoints Stimulation on Lung Complication After Abdominal Surgery
Brief Title: Dual Acupoints Stimulation Alleviates Pulmonary Complication
Acronym: DALAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Zhihong LU, Clinical Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJH-A-2016-10-10
Record Dates: First submitted 2017-07-10; First posted 2017-07-26 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pulmonary Complication; Postoperative Complications
Keywords: acupoint stimulation; elderly patients; postoperative pulmonary complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupoint stimulation (Experimental): Acupoint Zhongfu and Zusanli are stimulated by transcutaneous electrical stimulation
  Interventions: Device: acupoint stimulation
- no treatment (Sham Comparator): Electrodes are attached to Acupoint Zhongfu and Zusanli, but no stimulation is given
  Interventions: Device: no treatment

INTERVENTIONS:
Device: acupoint stimulation — Acupoint Zhongfu and Zusanli are stimulated through electrodes attached on the skin
  Other Names: transcutaneous electrical acupoint stimulation
  Arms: Acupoint stimulation
Device: no treatment — electrodes are attached, but no stimulation is given
  Other Names: control
  Arms: no treatment

SUMMARY:
Stimulation at acupoints could be of beneficial effects during the perioperative period. In this study the investigators tend to verify the effect of dual acupoints stimulation on pulmonary complications after abdominal surgery in aged patients.

DETAILED DESCRIPTION:
Postoperative pulmonary complications contributes to the high morbidity of aged patients. The incidence could be as high as 30~50% in those undergoing abdominal surgery. Stimulation at acupoints have been to alleviate inflammatory response,improve pain management and decrease consumption of opioids, indicating a beneficial effect on pulmonary complications. In this study the investigators tend to verify the effect of dual acupoints stimulation on pulmonary complications after abdominal surgery in aged patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed consented
* Scheduled for elective abdominal surgery under general anesthesia
* Age >=65 yrs

Exclusion Criteria:

* Patients with contraindications to transcutaneous electrical stimulation
* Patients with difficulty in communication that may confuse follow-up
* emergent surgeries
* Patients with pneumonia or needed ventilation before surgery
* Patients with history of pulmonary surgery
* Scheduled surgery involves thoracic manipulations
* Patients who attended clinical studies in the last 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12-10 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
incidence of pulmonary complications in 30d post-surgery | from end of surgery to Day 30 after surgery, totally 30 days
  incidence of pulmonary complications including pneumonia,atelectasis, pleural effusion and respiratory failure

SECONDARY OUTCOMES:
ICU admission after surgery | from end of surgery to Day 30 after surgery, commonly in 24h after surgery
  incidence of patients admitted to ICU unexpectedly
ICU stay after surgery | from admission to ICU to being discharged from ICU,averagely 2 days
  Time of patients stayed in ICU
Mortality in 30 days after surgery | from end of surgery to Day 30 after surgery, totally 30 days
  death of all causes
incidence of pulmonary complications in 3 days post-surgery | from end of surgery to Day 3 after surgery, totally 3 days
  incidence of pulmonary complications including pneumonia,atelectasis, pleural effusion and respiratory failure
Hospital stay after surgery | from end of surgery to being discharged from hospital,averagely 5 days
  Time of patients stayed in hospital after surgery
expense after surgery | from end of surgery to being discharged from hospital,averagely 5 days
  expense of patients after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, Prof., Study Chair — Air Force Military Medical University, China
Locations (3):
- China (3):
  - First Afiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - First Afiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rajamanickam T. Peri-operative care for the elderly. Anaesthesia. 2014 Mar;69(3):284-5. doi: 10.1111/anae.12616. No abstract available. PMID 24548361
- [Background] Guay J, Ochroch EA. Intraoperative use of low volume ventilation to decrease postoperative mortality, mechanical ventilation, lengths of stay and lung injury in patients without acute lung injury. Cochrane Database Syst Rev. 2015 Dec 7;(12):CD011151. doi: 10.1002/14651858.CD011151.pub2. PMID 26641378
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Moine P, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network investigators. Incidence of mortality and morbidity related to postoperative lung injury in patients who have undergone abdominal or thoracic surgery: a systematic review and meta-analysis. Lancet Respir Med. 2014 Dec;2(12):1007-15. doi: 10.1016/S2213-2600(14)70228-0. Epub 2014 Nov 13. PMID 25466352
- [Background] Lu Z, Dong H, Wang Q, Xiong L. Perioperative acupuncture modulation: more than anaesthesia. Br J Anaesth. 2015 Aug;115(2):183-93. doi: 10.1093/bja/aev227. PMID 26170347
- [Derived] Lu ZH, Dong HL, Huang-Fu JW, Fan XJ, Zhao WX, Min S, Zhang W, Liu MF, Wang YH, Wang LN, Xiong LZ. Effect of dual-acupoint and single-acupoint electric stimulation on postoperative outcomes in elderly patients subjected to gastrointestinal surgery: study protocol for a randomized controlled trial. Trials. 2018 Dec 4;19(1):669. doi: 10.1186/s13063-018-3052-2. PMID 30514358